CLINICAL TRIAL: NCT05527964
Title: The Influence of Specific Targeted Therapy on Subject and Family Quality of Life, Anxiety, Depression and Sleep Quality in Patients With Severe Refractory Atopic Dermatitis in the Czech Republic
Brief Title: A Study to Evaluate the Quality of Life of Male and Female Adult Patients With Severe Refractory Atopic Dermatitis Treated With Dupilumab in Czech Republic
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17350; U1111-1279-3216 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-08-22; First posted 2022-09-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with severe refractory atopic dermatitis: Patients eligible for Dupixent therapy of AD

SUMMARY:
Assessment of the relationship between treatment response (EASI75) and change in quality of life (EQ-5D) by week 24.

Description of the:

* Change in disease activity after 16 and 24 weeks
* Change in subject and family quality of life after 16 and 24 weeks
* Change in sleep quality after 16 and 24 weeks
* Change in anxiety after 16 and 24 weeks
* Change in depression after 16 and 24 weeks
* Safety and tolerability

DETAILED DESCRIPTION:
28 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for Dupixent therapy of AD according to the current SPC and reimbursement criteria given by the SUKL
* Signed informed consent
* 18 years and older (study questionnaires are validated for this age group). Patient is able to follow the prescribed regimen, routine follow-up visits and to fill the questionnaires

Exclusion Criteria:

- Patient not eligible for Dupixent therapy of AD according to the current SPC and reimbursement criteria given by the SUKL.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for Dupixent therapy of atopic dermatitis (AD) according to the current summary of product characteristics (SPC) and reimbursement criteria given by the State Institute for Drug Control (SUKL) in Czech Republic
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
The regression coefficient for at least 75% reduction in the Eczema Area and Severity Index score (EASI75) at week 24 adjusted to baseline characteristics predicting the change in EQ-5D utility | At Week 24

SECONDARY OUTCOMES:
Change in disease activity (Eczema Area and Severity Index (EASI) score) | At Week 16 and Week 24
Change in subject generic quality of life (European Quality of Life Five Dimension questionnaire (EQ-5D) utility) | At Week 16 and Week 24
Change in Dermatology Life Quality Index (DLQI score) | At Week 16 and Week 24
Change in Family Dermatology Life Quality Index (FDLQI score) | At Week 16
Change in sleep quality (Jenkins Sleep Evaluation Questionnaire (JSEQ) score) | At Week 16 and Week 24
Change in anxiety (Clinically Useful Anxiety Outcome Scale (CUXOS) score) | At Week 16 and Week 24
Change in depression (Clinically Useful Depression Outcome Scale (CUDOS) score) | At Week 16 and Week 24
Total number of adverse events | At Week 16 and Week 24
Number of serious adverse events (SAEs) | At Week 16 and Week 24
Number of non-serious adverse events (non-SAEs) | At Week 16 and Week 24
Total number of discontinuations | At Week 16 and Week 24
Reasons for discontinuations | At Week 16 and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site: Bulovka University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org